CLINICAL TRIAL: NCT04972305
Title: The Effect of the Prevention Program Developed for Injuries in Recreational Cyclists on Physical Performance and Physical Fitness Parameters
Brief Title: The Impact of the Prevention Program Developed for Injuries in Recreational Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, YUSUF ŞİNASİ KIRMACI, Pt, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YusufK
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Sports Physical Therapy
Keywords: recreational cyclist; exercise; physical fitness; sports performance
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Experimental): 12 weeks exercise programme, 3 days a week Bicycle ergonomics will be applied.
  Interventions: Other: Exercise and ergonomics
- Ergonomics group (Experimental): Bicycle ergonomics will be applied.
  Interventions: Other: Ergonomics
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Other: Exercise and ergonomics — 12 week exercise and fit bike
  Arms: Exercise group
Other: Ergonomics — Fit bike
  Arms: Ergonomics group

SUMMARY:
The aim of this study is to determine the effects of personal ergonomic adaptations of the bicycle on the bicycle performance parameters, together with the exercise program training created to prevent biomechanical problems that cause injuries in recreational cyclist.

DETAILED DESCRIPTION:
Considering the pandemic period we are living in, people are much more interested in health, sports and nature than they used to be. From this perspective, the interest in cycling, which can accommodate all of these features at the same time, is rapidly increasing. Individuals take bicycle rides in nature in their free time and make this activity a way of life. However, as in every physical activity, factors such as lack of knowledge in cycling, choosing the wrong bike and material, and not knowing the important basics of sports cause non-traumatic injuries in cyclists.

While transitioning from the sedentary life brought by the age of technology to the activity, the musculoskeletal systems of individuals are caught unprepared and even exposed to various traumas and biomechanical problems. Because the looping motion of the lower extremities while cycling occurs primarily in the sagittal plane, power imbalances can develop that affect a cyclist's susceptibility to injury elsewhere along the kinetic chain. The most common areas of overuse injury in cycling are the knee, lumbar spine, cervical spine, hip, Achilles tendon, wrists, and forearm.

ELIGIBILITY:
Inclusion Criteria:

* Recreational cycling for at least 1 year
* body mass index between 18.5-25 kg / m²
* Obtaining a written health report stating "there is no harm in using a bicycle"

Exclusion Criteria:

* History of fracture, trauma or surgery in the last 6 months
* have any systemic or neurological problems

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Body Composition | Change from Baseline at 12th weeks and 6th month
  Body fat percentage will be determined by skinfold measurement
Muscle strength | Change from Baseline at 12th weeks and 6th month
  It will be measured with "1 max rep" (1RM).
Flexibility | Change from Baseline at 12th weeks and 6th month
  It will be evaluated with sit-reach test and modified ober test.
Aerobic Capacity | Change from Baseline at 12th weeks and 6th month
  It will be evaluated by shuttle run.
Functional threshold power test (FTP) | Change from Baseline at 12th weeks and 6th month
  It is obtained by calculating the force applied while pedaling for 20 minutes.
Lactate threshold heart rate | Change from Baseline at 12th weeks and 6th month
  Average heart rate taken while pedaling for 20 minutes.
10-Mile Trial Test | Change from Baseline at 12th weeks and 6th month
  The time it takes to complete 10 miles in the fastest possible time is counted.
Critical Power test | Change from Baseline at 12th weeks and 6th month
  It is the estimation of the maximum effort that can be sustained for 3 minutes.
Muscle myotonometric properties | Change from Baseline at 12th weeks and 6th month
  It will be measured with myoton pro.
Balance | Change from Baseline at 12th weeks and 6th month
  It will be measured with Y balance test.

SECONDARY OUTCOMES:
Perceived pain | Change from Baseline at 12th weeks and 6th month
  It will be measured with McGill pain questionnaire
İnjury | Change from Baseline at 12th weeks and 6th month
  It will be measured with The Nordic musculoskeletal questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: GÜNSELİ USGU, Study Director — Hasan Kalyoncu University
Locations (1):
- Yusuf Şinasi Kirmaci, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No